CLINICAL TRIAL: NCT06847256
Title: Exploring a Common Genetic Risk Factor for Heat Stroke and Dehydration
Brief Title: Genetic Risk Factor for Heat Stroke
Status: Recruiting | Type: Observational
Sponsor: University of Iowa (Other)
Responsible Party: Principal Investigator, Aaron C. Miller, Research Assistant Professor, University of Iowa
Other Study IDs: 202308319
Record Dates: First submitted 2025-02-14; First posted 2025-02-26 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Carrier State; Heat Stroke; Dehydration
MeSH Terms: conditions — Heat Stroke; Dehydration

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- CF Carriers: Participants who have previously been genotyped as CF Carriers.
  Interventions: Procedure: Heat Challenge
- Controls: Participants who have previously been genotyped as controls and are age- and sex-matched to a CF Carrier.
  Interventions: Procedure: Heat Challenge

INTERVENTIONS:
Procedure: Heat Challenge — Participants will be asked to arrive well-hydrated and to refrain from exercise, alcohol, caffeine, and smoking for 24 hours prior to the visit. Height, weight, blood pressure, and body fat percentage will be measured. Blood (15.5 ml) and urine will be collected. Participants will wear a heart rate monitor and sit in a heat chamber at 62-63 degrees Celsius for 45 minutes. Heart rate will be measured continuously. Body temperature and a self-report of their comfort (1-4 scale) and thermosensation (1-7 scale) will be measured before the challenge, every 15 minutes during the challenge, and after the challenge. During the challenge, a sample of sweat will be collected to measure electrolyte loss. Participants will consume 16 ounces of water at their own pace during the 45 minutes. If they become too uncomfortable to continue or their body temperature rises above 39 degrees Celsius, the challenge will be stopped. All baseline measures except body fat percentage will be measured again.

SUMMARY:
The goal of this observational study is to examine the effect of the Cystic Fibrosis (CF) Carrier state on the risk for dehydration and other CF-specific fluid-and-electrolyte disorders in male and female adults.

The primary aim of the study is to estimate the risk of electrolyte disorders attributable to the CF carrier state in a genotyped cohort.

This will be accomplished with two smaller projects- Aim 1 and Aim 2.

Aim 1 will consist of 100 CF Carriers and 100 age- and sex-matched controls. Participants in this aim will be asked to complete a Participant Info and Temperature Survey consisting of questions about race, ethnicity, medical history, and how they experience heat.

Aim 2 will consist of a subset of 25 CF Carriers and 25 age- and sex-matched controls from Aim 1. Participants in this aim will be scheduled for a visit to complete a heat challenge. At this visit, they will also complete the Participant Info and Temperature Survey. They will also sit in a sauna at 62 - 63 degrees Celsius for 45 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Previously genotyped as a CF carrier or control
* Comfortable speaking/reading English

Exclusion Criteria:

* Previously genotyped as a CF patient
* Diagnosis of Type 1 or Type 2 diabetes
* History of heart attack, stroke, heart failure, or atherosclerosis
* Currently pregnant
* Currently taking beta blockers or diuretics
* Prisoner status
* Unable to provide own written informed consent

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Individuals who have previously been genotyped as CF Carriers or Controls.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-11-19 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Participant Scores for Temperature Sensitivity and Regulation Survey | Baseline
  Individual and composite scores for 5 components of the Temperature Sensitivity Survey (Heat- and Activity-Induced Autonomic Thermoregulation; Heat-Induced Behavioral Thermoregulation; Heat Perception; and Heat- and Activity-Induced Fatigue). For these 5 components, there are a total of 25 questions. All questions are on a 7-point scale, with the highest representing the most sensitive to heat and the lowest being the least sensitive. We will add up the scores for each question to arrive at a composite score for each component and the component scores will be added to arrive at a total score. Scores will be compared between groups.
Change in Weight | Up to 45 minutes
  Weight will be measured in kilograms pre- and post-heat challenge. We will compare change in weight between groups.
Change in Sodium Concentration | Up to 45 minutes
  Sodium concentration will be measured pre- and post-heat challenge by blood draw and urine sample. Sodium concentration will be compared between groups.
Change in Potassium Concentration | Up to 45 minutes
  Potassium concentration will be measured pre- and post-heat challenge by blood draw and urine sample. Potassium concentration will be compared between groups.
Concentration of Sweat Chloride | Up to 45 minutes
  Sweat chloride will be measured pre- and post-heat challenge by sweat collection. Sweat chloride will be compared between groups.
Final Score on Comfort Scale | Up to 45 minutes
  Participants will rate their level of comfort on a scale of 1-4 at the end of the heat challenge. Scores will be compared between groups.
Final Score on Thermosensation Scale | Up to 45 minutes
  Participants will rate their level of thermosensation on a scale of 1-7 at the end of the heat challenge. Scores will be compared between groups.

CONTACTS AND LOCATIONS:
Overall Officials: Aaron Miller, PhD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa Health Care, Iowa City, Iowa, United States